CLINICAL TRIAL: NCT04359433
Title: Evaluation the Effectiveness of Intermittent Anaerobic Exercise Among the Students With Cardiometabolic Risk
Brief Title: Intermittent Exercise Among Students
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issue
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IES-EKYY
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cardiometabolic Risk
Keywords: cardiometabolic; children; Waist to height ratio, WHtR; Intermittent Anaerobic Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (No Intervention): The participates in this group would provide normal health education of scientific and rational diet.
- Exercise intervention group (Experimental): Besides normal health education of scientific and rational diet，the participates in this group would be suggested to carry out an anaerobic exercise named Tabata.
  Interventions: Behavioral: Exercise programme

INTERVENTIONS:
Behavioral: Exercise programme — Exercise programme includes 8 anaerobic movements choosen from Tabata. This exercise programme workout is aimed at body fat reduction, and the structure is as follows:
  * 8 anerobic movements in 20 seconds is a set
  * Rest for 10 seconds before another set
  * Finish 4 sets every time, it shall take you 4 minutes
  * Do 4 sets 2 to 3 times a week
  Arms: Exercise intervention group

SUMMARY:
Evaluate the effectiveness of intermittency anaerobic exercise interventions among the students with high risk of cardiometabolic .

ELIGIBILITY:
Inclusion Criterias:

* Male: Waist-to-height ratio≥0.463
* Female： Waist-to-height ratio≥0.469
* Students with cardiometabolic risk factors include elevated BP, dyslipidaemia, elevated fasting blood glucose (FBG) and central obesity.

Exclusion Criterias:

* Participates with severe disease conditions include cardiac insufficiency, respiratory system relate diseases, immunodeficiency or severe malnutrition, ect
* Taking or having taken weight-loss drugs
* Participates unsuitable or improper to participate the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Abnormal of cardiometabolic risk related index | 3th month after enrollment
  Cardiometabolic risk related index includes fasting blood glucose, blood lipids, blood pressure and abdominal obesity.Cardiometabolic risk related index would be set to 1 as at least 2 indexs mentioned were abnormal while 0 for less than 2.

SECONDARY OUTCOMES:
Change of Waist-to-height ratio | Baseline, 12th months after enrollment
  Waist-to-height ratio is calculated by the formula ：Waist-to-height ratio=waistline (cm)/height(cm). All the participates' Waist-to-height ratio would be calculated at baseline and 12th months after enrollment. The change would be manifested in the situatuion of the difference.
Change of Body Mass Index | Baseline, 12th months after enrollment
  Body Mass Index is calculated by the formula ：Body Mass Index=weight(kg)/(height(cm))^2. All the participates' Body Mass Index would be calculated at baseline and 12th months after enrollment. The change would be manifested in the situatuion of the difference.
Change of hipline | Baseline, 12th months after enrollment
  All the participates' hipline would be measured at baseline and 12th months after enrollment. The change would be manifested in the situatuion of the difference.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Yan, PhD, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided